CLINICAL TRIAL: NCT02209883
Title: The Effects of Chronic Obstructive Pulmonary Disease on the Washout Time of Sevofluorane Anesthesia
Brief Title: The Effect of Sevofluorane on Wash-out Time in COPD
Acronym: washout
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Ilknur Suidiye, Assistant profesor, Duzce University
Other Study IDs: sevofluorane washout time COPD
Record Dates: First submitted 2014-07-22; First posted 2014-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia
Keywords: sevoflurane, anesthesia, washout time,COPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group normal: The patients which have not clinical diagnosis of chronic obstructive lung disease.
- Group COPD: The patients which have chronic obstructive lung disease in clinical evaluation

SUMMARY:
COPD (Chronic obstructive disease ) is a condition of respiratory system failure seen occasionally in elderly patients of society. Sevofluorane is a safe, volatile anesthetic used considerably widely all over the world. Because respiratory functions and gas exchange became impaired in COPD patients, the respiratory system excretion/washout of inhalational anesthetic agents can be affected. In our study we aimed to investigate if there is a relation between sevofluorane's washout time and the degree of COPD.

DETAILED DESCRIPTION:
Having approval by the Duzce University non-invasive clinical ethics committee and the written consent, the study was conducted by researchers among 60 American Society of Anesthesiologists (ASA) physical status 1 or 2 patients scheduled for orthopedic, urologic and lower limp surgery which performed under general anesthesia .We investigated patients who have normal pulmonary function and who have chronic obstructive pulmonary disease .We divided into two groups by via questioning and evaluating pulmonary function tests of patients.

The patients were 18-60 years old, with body mass index between 22-29. The exclusion criteria were:

1. Cardiac failure
2. Hepatic failure
3. Renal failure
4. Neurologic diseases
5. Endocrine diseases Study design Neither group received premedication. After being taken to the operating room all patients were monitored continuously throughout the study by standard ASA monitors. In addition to standard ASA monitors, inspired oxygen concentration (FiO2 ), inspired and expired concentration of sevofluorane, MAC levels of the patients were monitored.

Anesthesia was induced by propofol (2mg . kg-1), fentanyl (1,5-2 mcg. kg-1), rocuronium(0,6mg. kg-1) intravenously. General anesthesia was maintained by remifentanyl infusion(0,25-1 mcg.kg-1.min-1) and sevofluorane (1 MAC level corrected for the patients age). Fresh gas flow was 6 L. min-1 (50%-50% oxygen/air mixture). Patients were mechanically ventilated (Vt: 6-8 ml. kg-1 , frequency: 9-12 breath.min-1), adjusted to provide an end-tidal CO2 concentration of 35-40 mmHg and SpO2> %95 during anesthetic and surgical procedure.The patients non-invasive arterial tension and heart rate was maintain within normal limits. All data were recorded on each patient's observation charts.

At the end of the surgery, the sevofluorane vaporizer was turned off and the time taken for the sevofluorane concentration to decrease from 1 MAC to 0.3 MAC (MAC awake) and 0.1 MAC were recorded. The ratio of the fraction of inspired of sevoflurane and of expired concentration (Fexp) of sevofluorane at 1 MAC and Fexp of sevofluorane at 0.1 MAC were recorded. Mechanical ventilations of the patients were maintained until extubation and standardized according to ideal body weight. All patients extubated immediately after the patients were given reaction to the endotracheal tube. Remifetanyl infusion was maintained until 0.1 MAC level was reached.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists (ASA) physical status 1 or 2 patients
* orthopedic, urologic and lower limp surgery which performed under general anesthesia
* normal pulmonary function
* chronic obstructive pulmonary disease

Exclusion Criteria:

* Cardiac failure
* Hepatic failure
* Renal failure
* Neurologic diseases
* Endocrine diseases
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the study was conducted by reserchers among 60 American Society of Anesthesiologists (ASA) physical status 1 or 2 patients scheduled for orthopedic, urologic and lower limp surgery which performed under general anesthesia .We investigated patientes who have normal pulmonary function and who have chronic obstructive pulmonary disease .We divided into two groups by via questioning and evaluating pulmonary function tests of patients.
  The patients were 18-60 years old, with body mass index between 22-29
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
washout time | second
  The time in which sevoflurane MAC level decrease from 0.3 MAC to 0.1MAC and 0,1 MAC to extubation in the patients expiratory gases

SECONDARY OUTCOMES:
extubation time | seconds
  The time which sevoflurane MAC level decrease 1 MAC to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Suidiye Seker, Asist. prof., Study Director — Duzce University School of Medicine
Locations (1):
- Duzce Univercity Medical Fauculty, Düzce, Turkey (Türkiye)

REFERENCES:
- [Background] Adanir T, Atay A, Sencan A, Aksun M, Karahan N. Effect of cigarette smoking on the washout time of sevoflurane anesthesia. BMC Anesthesiol. 2010 Jun 22;10:8. doi: 10.1186/1471-2253-10-8. PMID 20569431
- See also: PMC full text — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2905413/